CLINICAL TRIAL: NCT01894412
Title: A Randomized, Double-blind, Single-dosing, Crossover Study to Compare the Safety and Pharmacokinetic Characteristics of HD203 25 mg With Those of Enbrel® Injection 25 mg After Subcutaneous Injection in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics of HD203 Liquid in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanwha Chemical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAGLE-I-13
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HD 203 (Experimental): prefilled syringe
  Interventions: Biological: Etanercept (Enbrel); Biological: HD203
- Enbrel (Active Comparator): prefilled syringe
  Interventions: Biological: Etanercept (Enbrel); Biological: HD203

INTERVENTIONS:
Biological: Etanercept (Enbrel)
Biological: HD203

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of HD203 liquid with those of etanercept (enbrel) prefilled injection after subcutaneous injection

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years of healthy volunteers

Exclusion Criteria:

* Subject who had been treated with Etanercept before

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | up to 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea